CLINICAL TRIAL: NCT07050732
Title: Immunogenicity and Safety of Multiple-Dose Adjuvanted RSVPreF3 (Arexvy®) Vaccination Among Immunocompromised Persons
Brief Title: Immunogenicity of RSVPreF3 Vaccine in Immunocompromised Persons
Acronym: STRIVE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00501702
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Syncytial Virus (RSV)
MeSH Terms: interventions — arexvy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: Arexvy + Placebo (Experimental): One dose of adjuvanted RSVPreF3 (Arexvy) at enrollment followed by placebo vaccine at Day 60 plus a re-vaccination Arexvy dose at 1 year (Day 365)
  Interventions: Biological: Arexvy (2 doses total); Other: Placebo
- Arm 2: Arexvy + Arexvy (Experimental): One dose of adjuvanted RSVPreF3 (Arexvy) at enrollment followed by a second dose of Arexvy at Day 60 plus a re-vaccination Arexvy dose at 1 year (Day 365)
  Interventions: Biological: Arexvy (3 doses total)
- Arm 3: Healthy Comparators (Experimental): One dose of adjuvanted RSVPreF3 (Arexvy) at enrollment
  Interventions: Biological: Arexvy (1 dose total)

INTERVENTIONS:
Biological: Arexvy (2 doses total) — Arexvy at enrollment, Arexvy at Day 365
  Other Names: adjuvanted RSVPreF3
  Arms: Arm 1: Arexvy + Placebo
Biological: Arexvy (3 doses total) — Arexvy at enrollment, Day 60, and Day 365
  Other Names: adjuvanted RSVPreF3
  Arms: Arm 2: Arexvy + Arexvy
Biological: Arexvy (1 dose total) — Arexvy at enrollment
  Other Names: adjuvanted RSVPreF3
  Arms: Arm 3: Healthy Comparators
Other: Placebo — Placebo vaccine at day 60
  Arms: Arm 1: Arexvy + Placebo

SUMMARY:
This clinical trial is being done to learn more about how well a vaccine (Arexvy®) for respiratory syncytial virus, also known as RSV, works in people with weakened immune systems. The main questions it aims to answer are:

* Does 1 or 2 doses of Arexvy work better in people with weakened immune systems?
* What medical problems do participants have after receiving Arexvy?

Participants with weakened immune systems will:

* Receive 3 study vaccines over the course of 1 year
* Keep a diary of symptoms for 7 days after each vaccine
* Have 3 in-person follow up study visits for checkups and tests over the course of 1.5 years
* Have 6 phone follow up study visits over the course of 1.5 years

DETAILED DESCRIPTION:
People with weakened immune systems will be randomized to either:

1. Receive one dose of Arexvy followed by a placebo vaccine (sterile saline) 60 days later, or
2. Receive one dose of Arexvy followed by another dose of Arexvy 60 days later

Both groups will also receive another dose of Arexvy 1 year after the first dose.

A small group of people without weakened immune systems will also be enrolled in the study. This group will receive one dose of Arexvy.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and provide informed consent
* Willing and able to comply with the requirements and restrictions in the protocol, including study visits and study-related procedures
* Medically stable in the opinion of the Investigator at the time of first study vaccination
* Life expectancy ≥ 365 days in the opinion of the Investigator at the time of first study vaccination
* Included in at least one of the groups below:

  1. Cellular therapy recipients (CTR):

     * Individuals ≥ 18 years of age at the time of first study vaccination
     * History of at least one of the following: i. Autologous stem cell transplant received more than 90 days prior to first study vaccination, ii. Allogeneic stem cell transplant received more than 90 days prior to first study vaccination, iii. Chimeric antigen receptor T cell (CAR-T) therapy received more than 90 days prior to first study vaccination
  2. Solid organ transplant recipients (SOTR):

     * Individuals ≥ 18 years of age at the time of first study vaccination
     * Received an ABO-compatible, single-organ type, solid organ transplant (lung, heart, kidney, liver) at least 90 days prior to first study vaccination, and are on at least 2 systemic immunosuppressive agents at time of first study vaccination
  3. Healthy comparator (HC):

     * Individuals ≥ 60 years of age at the time of first study vaccination or 50-59 years of age at the time of first study vaccination and at increased risk of severe RSV disease
     * No history of (a) or (b) above, and considered healthy or with chronic and stable medical conditions in the opinion of the Investigator, without immune compromise
* Participants of childbearing potential if practicing adequate contraception or abstinence from 1 month prior to first study vaccination and agree to continue adequate contraception or abstinence through at least 1 month after last study vaccination. All participants of childbearing potential must have a negative pregnancy test on the day of first study vaccination, prior to administration.

Exclusion Criteria:

* Known history of hypersensitivity to any vaccine or history of a life-threatening reaction to a vaccine
* Previous vaccination with any licensed or investigational RSV vaccine
* Acute or chronic clinically significant/unstable neurological disease (such as uncontrolled seizures, strokes, Guillain-Barré Syndrome (GBS)
* Vaccination with any inactivated, subunit, or split influenza vaccine or COVID-19 vaccine within 14 days prior to first study vaccination, or vaccination with any other licensed or investigational vaccine within 30 days prior to first study vaccination
* Receipt of investigational or approved monoclonal antibodies against RSV within 90 days prior to first study vaccination
* Moderate or severe acute illness/infection (in opinion of the Investigator) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of first study vaccination. A prospective participant should not be enrolled in the study until the condition has resolved or the febrile event has subsided.
* Any medical condition that in the opinion of the Investigator would make intramuscular injection unsafe
* Receipt of immunoglobulins or plasma products within 90 days prior to first study vaccination
* Receipt of B-cell depleting medications (e.g., Rituximab, ocrelizumab, ofatumumab, belimumab, epratuzumab, antithymocyte globulin) within 90 days prior to first study vaccination
* Currently pregnant or breastfeeding or planning to become pregnant, discontinue contraception, or breastfeed during the study period
* Any of the following:

  1. Cellular therapy recipients (CTR):

     * Graft-versus-host disease (GVHD) requiring systemic treatment with at least 0.5 mg/kg per day of prednisone or equivalent at time of first study vaccine
  2. Solid organ transplant recipients (SOTR):

     * History of any of the following within 90 days prior to first study vaccination: allograft rejection, post-transplant lymphoproliferative disease, treatment for either of these conditions
  3. Healthy comparator (HC):

     * Any confirmed/suspected immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive or cytotoxic therapy, based on medical history
* Any other conditions which, in the opinion of the Investigator, may pose additional risks from participation in the study, may interfere with the individual's ability to comply with study requirements or may impact the quality or interpretation of the data obtained from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Titer (GMT) (ED60 RSV A and B) | At 30 days post 1st and 2nd dose in Arm 1 and Arm 2
  Immune response elicited by adjuvanted RSVPreF3 (Arexvy) in immunocompromised adults as determined by titers of neutralizing antibody estimated dilution 60 (ED60) against RSV A and B
Immune response elicited by adjuvanted RSVPreF3 (Arexvy) in immunocompromised adults as determined by titers of neutralizing antibody ED60 against RSV A and B | At 30 days post 2nd dose (Arm 2) and 30 days post 1st dose (Arm 1)
  Mean Geometric Increase (MGI): Geometric mean of individual ratio of post-vaccine ED60 of RSV A and B over baseline titer (also called Geometric Mean Fold Rise [GMFR])

SECONDARY OUTCOMES:
Proportion of participants reporting reactions at injection site | Within 7 days of study vaccine administration
  Solicited local reactions including pain at injection site, erythema, and swelling
Proportion of participants reporting systemic events | Within 7 days of study vaccine administration
  Solicited systemic events including headache, fever, myalgia, arthralgia
Proportion of participants reporting adverse events | Through 30 days after each study vaccine administration
  Proportion of participants reporting adverse events
Adverse events of special interest | From enrollment to last study visit, approximately 18 months for Arms 1 and 2 and 12 months for Arm 3
  Proportion of participants reporting adverse events of special interest
Serious adverse events | Through 6 months following each study vaccine administration
  Proportion of participants reporting serious adverse events
Individual titers (ED60) for RSV-A and RSV-B #1 | 30 days post one year re-vaccination (Arm 1 and Arm 2)
  GMT
Individual titers (ED60) for RSV-A and RSV-B #2 | 30 days post 1st dose (Pooled Arm 1 and Arm 2; and Arm 3)
  GMT
Individual titers (ED60) for RSV-A and RSV-B #3 | 30 days post 1st dose (Pooled Arm 1 and Arm 2; and Arm 3)
  GMFR
Individual titers (ED60) for RSV-A and RSV-B #4 | 30 days post 2nd dose (Arm 2)
  GMFR
Individual titers (ED60) for RSV-A and RSV-B #5 | At 30 days after each study vaccine administration
  Seroresponse rate (% of participants with at least a 4-fold increase from baseline in RSV A and RSV B ED60)
Individual titers (ED60) for RSV-A and RSV-B #6 | At 30 days post a one year re-vaccination (Arm 1 and Arm 2)
  GMFR
Cell mediated immunity (RSV F specific CD4+ and CD8+ T cell response (T cells producing ≥ 2 cytokines, expressed as % of live CD3+)) #1 | At 30 days post 2nd dose (Arm 2) and 30 days post 1st dose (pooled Arm 1 and 2; and Arm 3)
  Median cell mediated immunity (CMI)
Cell mediated immunity (RSV F specific CD4+ and CD8+ T cell response (T cells producing ≥ 2 cytokines, expressed as % of live CD3+)) #2 | At 30 days post 1st dose (Pooled Arm 1 and Arm 2; and Arm 3)
  Median CMI
Cell mediated immunity (RSV F specific CD4+ and CD8+ T cell response (T cells producing ≥ 2 cytokines, expressed as % of live CD3+)) #3 | At 30 days post one year re-vaccination (Arm 1 and Arm 2)
  Median CMI

CONTACTS AND LOCATIONS:
Overall Officials: John Baddley, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No